CLINICAL TRIAL: NCT01877863
Title: The Effect of Intradialytic Exercise on the Functional Capacity of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr Jennifer MacRae, Principal Investigator, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-25253
Record Dates: First submitted 2013-05-27; First posted 2013-06-14 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: End Stage Kidney Disease
Keywords: intradialytic exercise; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intradialytic exercise (Experimental): baseline data prior to starting exercise program will be obtained and then compared to the data after 12 weeks of an intradialtyic biking program
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — 12 weeks of intradialytic biking at Borg intensity 3 - 4 for 15 to 60 minutes on each dialysis run
  Other Names: intradialytic exercise; intradialytic biking; biking on hemodialysis

SUMMARY:
The purpose of this study is to explore the impact of an intradialytic exercise program on functional capacity, aerobic capacity, strength, quality of life, depression, hospitalizations and intradialytic episodes of hypotension. The investigators would also like to look at the impact of exercise training over twelve weeks on hemoglobin levels as well as the clearance of potassium, phosphate and urea. Our hypothesis is that the above mentioned outcomes will positively improve over the twelve week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac and hemodynamic stability
* Absence of severe musculoskeletal impairment
* Increased musculoskeletal weakness
* Vital signs within normal range for exercise
* Desire/motivated to exercise
* Clearance from nephrologist and Kinesiologist

Exclusion Criteria:

* Compromised cardiac profiles
* Hemodynamic instability
* Severe bone disease
* Medical conditions which contraindicate exercise

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 12 weeks
  Functional capacity is measured by the DASI score which gives an estimated V02 peak in ml/min/kg. The difference between the mean score at baseline and 12 weeks will be determined.

SECONDARY OUTCOMES:
Aerobic capacity | 12 weeks
  Aerobic capacity is measured as a function of the DASI score
Strength | 12 weeks
  Strength is determined as bilateral hand grip strength (measured in kg) as well as by the 30 second sit to stand test(the number of repetitions achieved in 30 seconds). These measures are obtained at baseline and again at 12 weeks.
Quality of life | 12 weeks
  The KDQOL- SF36 will be used to measure the quality of life at baseline and again at 12 weeks.
Hospitalizations | 12 weeks
  The number and rate of hospitalizations will be determined prior to exercise start and during the 12 week exercise program. Length of stay is also tracked.
Hypotension | 12 weeks
  Intradialytic hypotension, defined as a drop in systolic blood pressure (SBP) of 20 mmHg for patients with pre-dialysis blood pressure > 100 mmHg or a drop in SBP of 10 mmHg for patients with pre-dialysis blood pressure < = 90 mmHg. IDH with patient symptoms and nursing interventions will be obtained as well.
Hemoglobin levels | 12 weeks
  The baseline hemoglobin and hemoglobin at 12 weeks will be tracked.
Potassium levels | 12 weeks
  The baseline potassium and potassium at 12 weeks as well as the K gradient (pre -dialysis - dialysate K level)will be monitored.
Urea removal | 12 weeks
  The baseline and 12 week pre and post dialysis urea levels will be monitored.
Phosphate levels | 12 weeks
  The baseline and 12 week pre-dialysis phosphate levels will be tracked.
Bioimpedance derived volume and body mass determinations | 12 weeks
  In a small subset of patients (n=10) the bioimpedance derived fluid compartments (ECF, ICF, E:I ratio) and fat free body mass will be determined at both baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer MacRae, Principal Investigator — University of Calgary
Locations (1):
- Northwest Dialysis Centre, Calgary, Alberta, Canada